CLINICAL TRIAL: NCT02974608
Title: Demographic Surveillance to Monitor Impact of Malaria on Pregnant Women in Ouelessebougou, Mali
Brief Title: Impact of Malaria on Pregnant Women in Ouelessebougou, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917018; 17-I-N018
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03-21

CONDITIONS: Malaria
Keywords: Placental; Fetal Loss; Observational; Antenatal; Infection; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children 0-10 years: Children living in selected villages surrounding the district of Ouelessebougou
- Pregnant Women + Newborns: Pregnant women of any age and their newborn children
- Women of Child Bearing Age Potential: Non-pregnant women of child-bearing age

SUMMARY:
Background:

Malaria is a serious disease. It is passed by infected mosquitoes. In many parts of Africa, malaria continues to be the main cause of death in young children and pregnant women. Researchers want to find out more about how malaria affects pregnant women and their babies.

Objectives:

To study the rate of miscarriage and stillbirth during the second and third trimesters among women in a certain district in Mali. To study rates of malaria infection over time among pregnant women and children in this area.

Eligibility:

Pregnant women of any age and pregnancy stage and their newborns. They must live in Ouelessebougou, Mali. Children up to 10 years old who live there.

Design:

Information about the study will be shared at community meetings, during visits to the health centers, and during census updates.

Participants will read and sign a consent form.

Pregnant women will be screened to see if they are eligible. They may have a urine test. They may have an ultrasound to date their pregnancy. Ultrasound uses sound waves to take pictures of the body.

Women will be enrolled in the study after they have their babies.

Participants may have a physical exam.

Some participants will provide a finger/heel prick blood sample.

Participants will complete a questionnaire. They will be asked about:

Medical history

Antimalarial and other interventions

Socioeconomic status

Their pregnancy

Previous pregnancies

Health of their newborn...

DETAILED DESCRIPTION:
Placental malaria (PM) leads to poor outcomes for pregnant women and their babies, and is caused by Plasmodium falciparum sequestration in the intervillous spaces of the placenta and ensuing inflammation. Severe maternal anemia, low birth weight (LBW) delivery and fetal loss are common sequelae. Malaria-related LBW alone is estimated to cause 62,000-363,000 infant deaths in Africa each year. To reduce poor pregnancy outcomes associated with malaria infection, WHO recommends monthly anti-malarial treatment with sulfadoxine pyrimethamine (SP) during the second and third trimester and the use of insecticide-treated bed nets. However, in East and Southern Africa, SP has lost its efficacy due to the spread of drug-resistant parasites. Therefore, an effective vaccine for PM is needed. Although the ideal vaccine will be given to adolescent girls prior to becoming pregnant, at this early stage of pregnancy malaria vaccine development, it is unknown if a boosting dose may be needed during pregnancy.

Before testing new interventions to improve pregnancy outcomes, it is important to obtain baseline information on pregnancy outcomes in the target population. In our recent longitudinal study of 1,885 pregnant women in Mali, in which women were closely followed during pregnancy (including malaria prevention and treatment), 2.9%, 2.4% and 6% of pregnancies ended in miscarriage, stillbirth, and preterm delivery, respectively.

The primary goal of the study is to assess pregnancy outcomes in women in the community with access to the WHO recommended standard of care. In the first part of the study, all women presenting for an antenatal visit at Ouelessebougou health centers will be recruited into the study. In the second part of the study, non-pregnant women will be enrolled and followed to capture data on pregnancy outcomes including early pregnancy losses. Pregnancy outcome information will be collected after the birth of the child or after pregnancy termination (i.e. miscarriage/stillbirth). Primary and secondary endpoints will be analyzed using appropriate statistical methods, including possible confounders, to determine the prevalence and factors associated with poor pregnancy outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

A study participant must satisfy the following criteria to be enrolled in this study:

1. Pregnant women and their newborn cohort: Pregnant women of any age and pregnancy stage and their newborns residing in the study area
2. women of child-bearing age cohort: women who are not under contraception or breastfeeding for less than 12 months and planning to become pregnant, and their newborn once they become pregnant
3. Children between the ages of 0-10 years residing in the study area
4. The study participant or parent/guardian understands the study and is able to provide informed consent for themselves and/or their child.

EXCLUSION CRITERIA:

1. Temporary residence in the study area
2. Conditions that in the judgment of the investigator could impair the ability of the participants to understand the study or comply with the study procedures.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population from which the cohorts will be selected live in selected villages surrounding the districts of Ouelessebougou, Mali
Sampling Method: Non-Probability Sample
Enrollment: 7691 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of malaria infection | Semi-annual
  Rates of malaria infections
Assess the rate of fetal loss during the 2nd and 3rd trimesters | Annual
  Rates of fetal losses

SECONDARY OUTCOMES:
Assess the prevalence rate of SP resistant parasites | Annual
  Rate of SP resistant parasites (in vivo and molecular markers)
Assess the rate of pre-term and low birth weight deliveries | Annual
  Number of pre-term deliveries, low birthweight deliveries, neonatal mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fried, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ouelessebougou Clinical Research Center (Malaria Research and Training Center), Bamako, Mali